CLINICAL TRIAL: NCT05201807
Title: Evaluation of Marketed Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-6483
Record Dates: First submitted 2022-01-10; First posted 2022-01-21 (Actual); Results first posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TEST Lens (Experimental): Eligible subjects who are habitual soft contact lens wearers will be given the TEST Lens for the duration of the study.
  Interventions: Device: Dailies Total 1 (DT1)

INTERVENTIONS:
Device: Dailies Total 1 (DT1) — TEST Lens

SUMMARY:
This is a bilateral, 2-week dispensing, non-randomized, controlled, single-masked, single-arm study to evaluate overall vision and comfort

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 39 (inclusive) years of age at the time of screening.
4. By self-report, habitually wear spherical soft silicone hydrogel contact lenses in both eyes in a daily wear or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 5 days per week during the past 30 days.
5. Possess a wearable pair of spectacles that provide correction for distance vision.
6. The spherical equivalent of the subject's vertex-corrected distance refraction must be between -1.00 and -6.00 DS (inclusive) in each eye.
7. The magnitude of the cylindrical component of the subject's vertex-corrected distance refraction must be between 0.00 and 1.00 DC (inclusive) in each eye.
8. The best corrected, monocular, distance visual acuity must be 20/25or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Be currently pregnant or lactating.
2. Be currently using any ocular medications or have any ocular infection of any type.
3. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that the investigator believes might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
4. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
5. Be currently wearing monovision or multifocal contact lenses.
6. Be currently wearing lenses in an extended wear modality.
7. Have participated in a contact lens or lens care product clinical trial within 14 days prior to study enrollment.
8. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
9. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that the investigator believes might contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis). (Specify method of determination if needed).
10. Have a history of strabismus or amblyopia.
11. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
12. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (4):
- United States (4):
  - VisualEyes, Roswell, Georgia
  - Professional Vision Care Inc. - Westerville, Westerville, Ohio
  - Tyler Eye Associates, Tyler, Texas
  - William J. Bogus O.D., Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 80 subjects were enrolled in this study. The 80 enrolled subjects met all eligibility criteria and were dispensed at least one study lens. Of those dispensed, 78 subjects completed the study while 2 subjects were discontinued.
Groups:
- DT1 (Delefilcon A): Subjects that wore the DT1 lens during the study.
Period: Overall Study
Arm/Group | DT1 (Delefilcon A)
Started | 80
Completed | 78
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — COVID-19 Related | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Arm/Group | DT1 (Delefilcon A)
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.5 (5.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 34
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 6
  Black or African American | 7
  White | 67
Region of Enrollment [Number; unit: Participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Overall Quality of Vision Score
Description: Overall quality of vision score was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE vision score for each lens type was reported.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DT1 (Delefilcon A)
Number analyzed (Participants) | 78
Units on a scale | 56.9 (25.18)

2. Primary Outcome: Overall Quality of Comfort Score
Description: Overall quality of comfort score was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE comfort score for each lens type was reported.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DT1 (Delefilcon A)
Number analyzed (Participants) | 78
Units on a scale | 56.3 (29.21)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; The study duration for each subject was approximately 2 weeks.
Arm/Group | DT1 (Delefilcon A)
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT05201807/Prot_SAP_000.pdf